CLINICAL TRIAL: NCT00791700
Title: AN OPEN-LABEL, MULTICENTER, MULTIPLE-DOSE PHARMACOKINETIC, SAFETY AND EFFICACY TRIAL OF MARAVIROC IN COMBINATION WITH OPTIMIZED BACKGROUND THERAPY FOR THE TREATMENT OF ANTIRETROVIRAL-EXPERIENCED CCR5-TROPIC HIV-1 INFECTED CHILDREN 2 - <18 YEARS OF AGE
Brief Title: An Open Label Pharmacokinetic, Safety And Efficacy Study Of Maraviroc In Combination With Background Therapy For The Treatment Of HIV-1 Infected, CCR5 -Tropic Children
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ViiV Healthcare (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4001031; 2008-006873-33 (EudraCT Number)
Record Dates: First submitted 2008-11-12; First posted 2008-11-14 (Estimated); Results first posted 2016-02-25 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Human Immunodeficiency Virus
Keywords: Open label pharmacokinetic safety and efficacy in HIV-1 infected pediatrics
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Maraviroc (Experimental): Subjects will be stratified by age and formulation into one of the following cohorts:
  Cohort 1: ≥2-<6 years of age, maraviroc liquid formulation; Cohort 2: ≥6-<12 years of age, maraviroc tablet formulation; Cohort 3: ≥6-<12 years of age, maraviroc liquid formulation and Cohort 4: ≥12-<18 years of age, maraviroc tablet formulation.
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — Maraviroc will be administered twice daily either as a liquid or tablet formulation, depending on the age of the subject. The dosage administered will be dependent upon the subject's body surface area as well as the background therapy.
  Other Names: Selzentry

SUMMARY:
The primary purpose of this study is to determine the pharmacokinetic properties (what the body does to maraviroc) and to determine a suitable dosing schedule of maraviroc in HIV-1 infected children and adolescents. This study will also determine whether maraviroc is safe to use in children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 2-18 years of age, treatment experienced for 6 months or longer with at least 2 ARV drug classes, with HIV-1 RNA ≥1,000 copies/mL

Exclusion Criteria:

* X4- or dual/mixed-tropic virus detected by the Trofile™ viral tropism assay
* Concomitant therapy with other investigational agents (other than experimental ARV agents available through pre-approval access programs)
* Known ≥Grade 3 of any of the following laboratory tests at Screening or within 30 days prior to Baseline Visit: Neutrophil count, hemoglobin, platelets, AST, ALT, and creatinine, lipase;
* Total bilirubin ≥Grade 3, unless ALL of the following are true: Current regimen includes atazanavir; ALT/AST < 2.5 X ULN; No symptoms other than jaundice or icterus.
* Other laboratory values ≥Grade 3, must be reviewed by Pfizer.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 103 (Actual)
Dates: Start 2009-04-22 (Actual); Primary Completion 2015-04-14 (Actual); Study Completion 2023-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (41):
- United States (18):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Rainbow Center at University of Florida Health, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Grady Health System, IDP, Atlanta, Georgia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Pediatric Infectious Disease Clinic, Jackson, Mississippi
  - Batson Specialty Clinic, Jackson, Mississippi
  - University of Mississippi, Jackson, Mississippi
  - Cincinnati Center for Clinical Research, Cincinnati, Ohio
  - Children's Medical Center of Dallas, Dallas, Texas
  - Children's Memorial Hermann Hospital, Houston, Texas
  - UT Physician, Houston, Texas
  - VCU Health System Clinical Research Services, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Brazil (2):
  - Instituto de Infectologia Emilio Ribas, São Paulo, São Paulo
  - Condomínio Edifício Parque Paulista, São Paulo
- Italy (4):
  - Clinica Pediatrica Azienda Ospedaliera di Padova, Padua
  - Farmacia Interna, Padua
  - IRCCS Ospedale Pediatrico Bambino Gesu, Roma
  - Struttura Complessa a Direzione Universitaria Immunologia, Reumatologia e Malattie Infettive, Torino
- Hospital Infantil de Mexico Federico Gomez, Mexico City, Mexico City, Mexico
- Portugal (4):
  - Centro Hospitalar Universitario do Algarve, EPE, Faro
  - Centro Hospitalar de Lisboa Central, EPE, Lisbon
  - Centro Hospitalar de Lisboa Norte, EPE, Lisbon
  - Hospital S. João, E.P.E, Porto
- Hospital San Juan Research Unit, San Juan, PR, Puerto Rico
- South Africa (5):
  - Iatros International, Bloemfontein, Free State
  - Lakeview Hospital, Benoni, Gauteng
  - Dr George Mukhari Hospital, Ga-Rankuwa, Gauteng
  - Dr. Jan Fourie Medical Centre, Dundee, KwaZulu-Natal
  - Embassy Drive Medical Center, Pretoria
- Spain (2):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Barcelona, Spain
  - Hospital Universitario 12 de Octubre, Madrid
- Thailand (4):
  - Department of Pediatric, Faculty of Medicine, Khon Kaen University, Muang, Changwat Khon Kaen
  - Department of Pediatrics, Faculty of Medicine, Chiang Mai University, Muang, Chiang Mai
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT),, Bangkok
  - Department of Pediatrics, Faculty of Medicine, Siriraj Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4001031&StudyName=An%20Open%20Label%20Pharmacokinetic%2C%20Safety%20And%20Efficacy%20Study%20Of%20Maraviroc%20In%20Combination%20With%20Background%20Therapy%20For%20The%20Treatment%20Of%20HIV-

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This open-label, multicenter, multiple dose pharmacokinetic, safety and efficacy study at 24 sites in 8 countries.
Pre-assignment Details: The participants were HIV-1 infected treatment-experienced children and adolescents who were failing current antiretroviral (ARV) therapy or have failed their most recent ARV regimen, defined by plasma HIV-1 RNA>=1000 copies/mL, were infected with only R5 HIV-1, and have ARV experience/intolerance of 6 months with at least 2 ARV drug classes.
Groups:
- >=2 - <6 Years of Age, MVC Liquid Formulation: In Cohort 1, Participants aged >= 2 to < 6 years, received MVC liquid formulation (20 milligram per milliliter [mg/mL]).
- >=6 - <12 Years of Age, MVC Tablet Formulation: In Cohort 2, Participants aged >=6 to <12 years, received MVC tablet formulation (25 milligram [mg], 75 mg, 150 mg).
- >=6 - <12 Years of Age, MVC Liquid Formulation: In Cohort 3, Participants aged >=6 to <12 years, received MVC liquid formulation (20 mg/mL).
- >=12 - <18 Years of Age, MVC Tablet Formulation: In Cohort 4, Participants aged >=12 to <18 years, received MVC tablet formulation (25 mg, 75 mg, 150 mg).
Period: Overall Study
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Started | 16 | 31 | 13 | 43
Completed | 10 | 20 | 7 | 13
Not Completed | 6 | 11 | 6 | 30
Not completed — Insufficient clinical response | 1 | 4 | 1 | 8
Not completed — No longer willing to participate | 1 | 1 | 0 | 8
Not completed — Non-compliance with study treatment | 0 | 2 | 0 | 4
Not completed — Withdrawn due to pregnancy | 0 | 0 | 0 | 1
Not completed — Other | 0 | 1 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 4 | 3 | 4 | 6
Not completed — Adverse Event | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consisted of all participants who received at least 1 dose of study drug.
Groups:
- >=2 - <6 Years of Age, MVC Liquid Formulation: In Cohort 1, Participants aged >= 2 to < 6 years, received MVC liquid formulation (20 mg/mL).
- >=6 - <12 Years of Age, MVC Tablet Formulation: In Cohort 2, Participants aged >=6 to <12 years, received MVC tablet formulation (25 mg, 75 mg, 150 mg).
- Total: Total of all reporting groups
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation | Total
Number analyzed (Participants) | 16 | 31 | 13 | 43 | 103
Age, Continuous [Mean (Standard Deviation); unit: Years] | 3.4 (0.9) | 9.1 (1.7) | 8.9 (2.0) | 14.0 (1.6) | 10.3 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 16 | 6 | 27 | 54
  Male | 11 | 15 | 7 | 16 | 49

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic(PK): Maraviroc PK Parameter, Average Plasma Concentration (Cavg), Trough Concentration(Cmin), Maximum Plasma Concentration (Cmax)
Description: Cavg: calculated as area under the curve divided by a dosing interval of 12 hours. Cmin: directly observed plasma concentration prior to the next dose. Geometric Coefficient of Variation is defined as the geometric standard deviation to the power of the reciprocal of the geometric mean.
Time Frame: Week 2 and Week 48 (0, 1, 2, 4, 6, 8, 12 hours post-dose)
Population: PK analysis set consisted of all enrolled participants who had at least one PK sample with a dosing history. "Number analyzed": participants evaluable at specified time points for this measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 12 | 11 | 10 | 17
nanogram per milliliter (ng/mL)
  Cavg-Week2 | 237.34 (63) | 260.65 (43) | 264.45 (62) | 239.85 (67)
  Cavg-Week 48: number analyzed (Participants) | 9 | 8 | 8 | 12
  Cavg-Week 48 | 163.73 (146) | 289.69 (50) | 168.62 (117) | 199.12 (78)
  Cmax-Week2 | 581.47 (69) | 546.80 (51) | 444.37 (61) | 530.80 (62)
  Cmax-Week 48: number analyzed (Participants) | 9 | 8 | 8 | 12
  Cmax-Week 48 | 334.68 (156) | 593.68 (25) | 284.96 (128) | 423.32 (48)
  Cmin-Week2 | 18.97 (202208) | 100.02 (39) | 115.84 (90) | 56.17 (145)
  Cmin-Week 48: number analyzed (Participants) | 9 | 8 | 8 | 12
  Cmin-Week 48 | 48.11 (180) | 82.21 (120) | 60.03 (245) | 66.51 (140)

2. Primary Outcome: Area Under the Curve at Steady State (AUCtau)
Description: AUCtau is the area under the plasma concentration time curve (AUC) at steady state from time zero (pre-dose) to end of dosing interval (tau), here dosing interval is 12 hours.
Time Frame: Week 2 and Week 48 (0, 1, 2, 4, 6, 8, 12 hours post-dose)
Population: PK analysis set consisted of all enrolled participants who had at least one PK sample with a dosing history. "Number analyzed" signifies participants evaluable at specified time points for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 12 | 11 | 10 | 17
ng*hr/mL
  AUCtau - Week 2 | 2848.1 (63) | 3127.7 (43) | 3173.4 (62) | 2878.2 (67)
  AUCtau - Week 48: number analyzed (Participants) | 9 | 8 | 8 | 12
  AUCtau - Week 48 | 1964.7 (146) | 3476.3 (50) | 2023.5 (117) | 2389.4 (78)

3. Primary Outcome: Time to Reach Maximum Plasma Concentration (Tmax)
Time Frame: Week 2 and Week 48 (0, 1, 2, 4, 6, 8, 12 hours post-dose)
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 12 | 11 | 10 | 17
hour
  Tmax - Week 2 | 2.000 [0.97 to 6.00] | 4.000 [0.75 to 6.00] | 2.000 [1.00 to 4.00] | 2.000 [1.00 to 4.00]
  Tmax - Week 48: number analyzed (Participants) | 9 | 8 | 8 | 12
  Tmax - Week 48 | 2.000 [0.00 to 6.03] | 2.000 [1.00 to 8.00] | 3.000 [0.00 to 6.00] | 2.000 [1.00 to 4.00]

4. Primary Outcome: Incidence and Severity of Grade 3 and Grade 4 Treatment-Emergent Adverse Events(AEs) (All Causality)
Description: Incidence is reported in terms of number of events of AEs. The investigator used the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric AEs as follows: Grade 1= Symptoms causing no or minimal interference with usual social and functional activities; Grade 2= Symptoms causing greater than minimal interference with usual social and functional activities; Grade 3= Symptoms causing inability to perform usual social and functional activities; Grade 4= Symptoms causing inability to perform basic self-care functions or medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death. Data have been reported in the measure for Grade 3 and 4 as per system organ class and preferred term.
Time Frame: Baseline up to 5 years
Population: Safety analysis was performed on all participants who received at least 1 dose of study drug.
Measure: Number; unit: events
Groups:
- Cohort 1 (Grade 3): In Cohort 1, Participants aged >= 2 to < 6 years, received MVC liquid formulation (20 mg/mL).
- Cohort 1 (Grade 4): In cohort 1, Participants aged >= 2 to < 6 years, received MVC liquid formulation (20mg/mL).
- Cohort 2 (Grade 3); Cohort 2 (Grade 4): In Cohort 2, Participants aged >=6 to <12 years, received MVC tablet formulation (25 mg, 75 mg, 150 mg).
- Cohort 3 (Grade 3); Cohort 3 (Grade 4): In Cohort 3, Participants aged >=6 to <12 years, received MVC liquid formulation (20 mg/mL).
- Cohort 4 (Grade 3); Cohort 4 (Grade 4): In Cohort 4, Participants aged >=12 to <18 years, received MVC tablet formulation (25 mg, 75 mg, 150 mg).
Arm/Group | Cohort 1 (Grade 3) | Cohort 1 (Grade 4) | Cohort 2 (Grade 3) | Cohort 2 (Grade 4) | Cohort 3 (Grade 3) | Cohort 3 (Grade 4) | Cohort 4 (Grade 3) | Cohort 4 (Grade 4)
Number analyzed (Participants) | 16 | 16 | 31 | 31 | 13 | 13 | 43 | 43
events
  Gastrointestinal disorders - Vomiting | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Hepat. disorders - Drug-induced liver injury | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Infections and infestations - H1N1 influenza | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Infections and infestations - Pneumonia | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Investigations - Lipase increased | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Pyschiatric disorder - Bipolar disorder | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Gastrointestinal disorders - Gastritis | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Investigations - Hepatic enzyme abnormal | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Investigations - Transaminases increased | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Pyschiatric disorder - Aggression | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Blood and lymphatic system disorders - Anaemia | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Infections and infestations - Meningitis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Infections and infestations -Otitis media | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Treatment Discontinuation: Secondary Reasons- Serious Adverse Event (SAE) Related to Study Drug
Description: The primary reason for a participant discontinuing from study drug or the clinical study was recorded in the source documents as well as the case report form. A discontinuation had to be reported immediately to the study medical monitor or his/her designated representative if it was due to an SAE and was considered as a secondary reason.
Time Frame: Baseline up to 5 years
Population: Safety analysis was performed on all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 16 | 31 | 13 | 43
participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA <400 Copies/mL Through Week 48 Using Missing, Discontinuation = Failure (MD=F) Approach
Description: The proportion of participants who achieved HIV-1 RNA <400 copies/mL at week 24 or 48 was assessed according to Food and Drug Administration's (FDA's) Missing, Switch, Discontinuation'=Failure (MSDF) Snapshot algorithm. The algorithm uses the plasma HIV-1 RNA in the Week 24 or 48 visit window, follows the "virology-first principle" and considers a participant who has a missing plasma HIV-1 RNA, or switches to prohibited ARV regimen or discontinues from the study or study drug for any reason, or dies, as a failure.
Time Frame: Week 24 and Week 48 post-treatment
Population: The FAS consisted of all participants who receive at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 16 | 31 | 13 | 43
percentage of participants
  Week 24 | 68.8 | 90.3 | 69.2 | 62.8
  Week 48 | 75.0 | 77.4 | 69.2 | 51.2

7. Secondary Outcome: Percentage of Participants With HIV-1 RNA <48 Copies/mL Through Week 48 Using Missing, Discontinuation = Failure (MD=F)Approach
Description: The proportion of participants who achieved HIV-1 RNA <48 copies/mL at week 24 or 48 was assessed according to Food and Drug Administration's (FDA's) Missing, Switch, Discontinuation'=Failure (MSDF) Snapshot algorithm. The algorithm uses the plasma HIV-1 RNA in the Week 24 or 48 visit window, follows the "virology-first principle" and considers a participant who has a missing plasma HIV-1 RNA, or switches to prohibited ARV regimen or discontinues from the study or study drug for any reason, or dies, as a failure.
Time Frame: Week 24 and Week 48 post-treatment
Population: The FAS consisted of all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 16 | 31 | 13 | 43
percentage of participants
  Week 24 | 18.75 | 64.5 | 61.5 | 48.8
  Week 48 | 50.0 | 54.8 | 53.8 | 39.5

8. Secondary Outcome: Percentage of Participants With HIV-1 RNA Levels <400 Copies/mL at Weeks 24 and 48 Using Missing, Discontinuation = Failure (MD=F)Approach
Description: Participants who have been discontinued from the study, have been lost to follow-up, or have missing HIV-1 RNA data prior to the time point of interest were considered to have HIV-1 RNA levels > lower limit of quantification (LLOQ) . This referred to as [non-completer = failure; NC=F] or [missing, discontinuation = failure; MD=F].
Time Frame: Week 24 and Week 48 post-treatment
Population: The FAS consisted of all participants who received at least 1 dose of study drug. "Overall Number of Participants Analyzed" signifies the number of participants evaluable for this measure."Number analyzed" signifies participants evaluable at specified time points for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 12 | 27 | 9 | 27
Percentage of participants
  Week 24: number analyzed (Participants) | 10 | 27 | 9 | 27
  Week 24 | 62.5 [38.8 to 86.2] | 87.10 [75.3 to 98.9] | 69.2 [44.1 to 94.3] | 62.8 [48.3 to 77.2]
  Week 48: number analyzed (Participants) | 12 | 23 | 9 | 22
  Week 48 | 75.0 [53.8 to 96.2] | 74.2 [58.8 to 89.6] | 69.2 [44.1 to 94.3] | 51.2 [36.2 to 66.1]

9. Secondary Outcome: Percentage of Participants With HIV-1 RNA Levels < 48 Copies/mL at Weeks 24 and 48 Using MD=F Approach
Description: Participants who have been discontinued from the study, have been lost to follow-up, or have missing HIV-1 RNA data prior to the time point of interest were considered to have HIV-1 RNA levels > lower limit of quantification (LLOQ) . This referred as [non-completer = failure; NC=F] or [missing, discontinuation = failure; MD=F].
Time Frame: Week 24 and Week 48 post-treatment
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 8 | 20 | 8 | 21
Percentage of participants
  Week 24: number analyzed (Participants) | 3 | 20 | 8 | 21
  Week 24 | 18.8 [0.0 to 37.9] | 64.5 [47.7 to 81.4] | 61.5 [35.1 to 89.0] | 48.8 [33.9 to 63.8]
  Week 48: number analyzed (Participants) | 8 | 16 | 8 | 17
  Week 48 | 50.0 [25.5 to 74.5] | 54.8 [34.0 to 69.2] | 53.8 [35.1 to 89.0] | 39.5 [24.9 to 54.2]

10. Secondary Outcome: Percentage of Participants With HIV-1 RNA <400 Copies/mL and <48 Copies/mL Using the Time to Loss of Virologic Response Algorithm (TLOVR) at Week 48
Description: TLOVR is defined as the time from first dose of study medication (Day 1) until the time of virologic failure using the a TLOVR algorithm.
Time Frame: Week 48
Population: The FAS consisted of all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 16 | 31 | 13 | 43
Percentage of participants
  <400 copies/mL; TLOVR Responder | 62.5 | 74.2 | 69.2 | 48.8
  <48 copies/mL; TLOVR Responder | 43.8 | 54.8 | 46.2 | 44.2

11. Secondary Outcome: Percentage of Participants With >= 1.0 log10 Reduction in HIV-1RNA Concentration From Baseline to Week 24 and Week 48
Description: Percentage of participants with at least a 1.0 log10 reduction in HIV-1 RNA from baseline to Week 24 and Week 48 were tabulated.
Time Frame: Baseline to Week 24, Week 48 post-treatment
Population: The FAS consisted of all participants who received at least 1 dose of study drug. Last Observation Carried Forward (LOCF) was used to impute missing values.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 16 | 31 | 13 | 43
percentage of participants
  Baseline to Week 24 | 92.3 [77.8 to 106.8] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 93.1 [83.9 to 102.3]
  Baseline to Week 48 | 100.0 [100.0 to 100.0] | 96.2 [88.8 to 103.6] | 100.0 [100.0 to 100.0] | 88.0 [75.3 to 100.7]

12. Secondary Outcome: Change From Baseline in HIV-1 RNA (Original)
Description: Plasma HIV-1 RNA was determined using the Roche COBAS AmpliPrep/COBAS TaqMan HIV-1 Test (lower limit of quantification [LLOQ] <48 copies/mL). Blood samples were taken at the time points indicated in the participant evaluation schedule. Screening HIV-1 RNA >1000 copies/ml was used to determine eligibility for the study.
Time Frame: Baseline, Week 24, Week 48 post-treatment
Population: The FAS consisted of all participants who received at least 1 dose of study drug. LOCF was used to impute missing values. "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: copies/mL
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 15 | 31 | 12 | 39
copies/mL
  Change from Baseline - Original - Week 24 | -271974.6 (391843.59) | -38764.0 (63688.93) | -58081.0 (79720.33) | -57325.7 (172108.62)
  Change from Baseline - Original - Week 48 | -267834.2 (378896.88) | -34787.7 (60222.60) | -56351.7 (76231.03) | -55321.1 (173840.55)

13. Secondary Outcome: Change From Baseline in HIV-1 RNA (Log10 Copies/mL)
Description: as for outcome 12
Time Frame: Baseline, Week 24, Week 48 post-treatment
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Log10 Copies/mL
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 15 | 31 | 12 | 39
Log10 Copies/mL
  Change from Baseline - Log10 - Week 24 | -2.4853 (1.1421) | -2.2324 (0.8668) | -2.1756 (1.1854) | -1.6482 (1.3806)
  Change from Baseline - Log10 - Week 48 | -2.5831 (1.2148) | -1.9579 (1.0861) | -2.0549 (1.2125) | -1.4591 (1.4477)

14. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4+) Cell Count at Weeks 24 and 48
Description: Change from baseline in CD4 cell count to Week 24 and Week 48 were tabulated in aggregated and broken down by age cohort using summary statistics.
Time Frame: Baseline, Week 24, Week 48 post-treatment
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 15 | 30 | 12 | 39
cells/mm^3
  Week 24 | 232.7 (381.6) | 355.8 (294.0) | 213.9 (166.4) | 173.6 (203.6)
  Week 48 | 275.9 (363.4) | 362.7 (373.5) | 167.3 (150.9) | 168.6 (211.0)

15. Secondary Outcome: Change From Baseline in Percentage (%) of CD4+ Cells at Weeks 24 and 48
Description: Change from baseline in CD4 % to Week 24 and Week 48 were tabulated in aggregated and broken down by age cohort using summary statistics.
Time Frame: Baseline, Week 24 and Week 48 post-treatment
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: percentage of CD4+ cells
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 15 | 31 | 12 | 39
percentage of CD4+ cells
  Week 24 | 7.3 (5.0) | 3.8 (7.4) | 3.5 (4.0) | 3.8 (6.1)
  Week 48 | 7.5 (7.6) | 6.0 (6.8) | 2.5 (4.2) | 4.6 (6.5)

16. Secondary Outcome: Number of Participants With Protocol Defined Virologic Failure
Description: The occurrence of any one of the following criteria would constitute Virologic failure: Criteria A=Decrease from Baseline plasma HIV-1 RNA <1 log10 and plasma HIV-1 RNA >400 copies/mL starting at Week 12 and confirmed at consecutive Week 16; Criteria B=Decrease from Baseline plasma HIV-1 RNA <2.0 log10 and plasma HIV-1 RNA >400 copies/mL at Week 24 OR plasma HIV-1 RNA >10,000 copies/mL on and after Week 24, and confirmed within 14 to 21 days; Criteria C=Increase from nadir plasma HIV-1 RNA of >=1 log10 (>=1,000 copies/mL if nadir plasma HIV-1 RNA <48 copies/mL) at any time, and confirmed within 14 to 21 days.
Time Frame: Week 48
Population: The FAS consisted of all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 16 | 31 | 13 | 43
participants
  Criteria A | 0 | 2 | 1 | 5
  Criteria B | 0 | 0 | 0 | 0
  Criteria C | 3 | 3 | 2 | 8

17. Secondary Outcome: Number of Participants With Viral Tropism Between Screening and Confirmed Protocol Defined Virologic Failure (PDVF) Prior to Week 48
Description: Virus tropism was determined using the Monogram Biosciences Trofile™ viral tropism assay. Change in detected tropism from screening to the time of failure prior to Week 48 was reported. X4=CXCR4 tropic virus; R5=CCR5-tropic virus; X4=CXCR4-tropic virus. Number of participants as per tropism to respective virus has been reported.
Time Frame: Screening to Week 48
Population: Participants who experienced confirmed PDVF through Week 48 with sufficient plasma HIV-1 RNA for virology analysis while receiving MVC. One participant was excluded from summary tables as classified as MSDF response; one participant was analyzed after stopping treatment.
Measure: Number; unit: participants
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 3 | 4 | 3 | 13
participants
  With valid on-treatment results | 2 | 4 | 3 | 11
  Tropism at Confirmed PDVF R5 | 2 | 3 | 2 | 9
  Tropism at Confirmed PDVF DM | 0 | 1 | 1 | 2
  Tropism at Confirmed PDVF X4 | 0 | 0 | 0 | 0
  Tropism at Confirmed PDVF Not Reportable | 1 | 0 | 0 | 1

18. Secondary Outcome: Number of Participants With Emergence of Reverse Transcriptase Inhibitor (RTI) and Protease Inhibitor (PI) Resistance Associated Mutations (RAMs) Between Screening and On-Treatment Confirmed PDVF
Description: Phenotypic and genotypic susceptibility to reverse transcriptase and protease inhibitors was evaluated at screening using the Monogram Biosciences PhenoSense™ GT (PSGT) assay. Samples from a confirmatory PDVF visit or early termination of MVC were planned to be analyzed if the plasma HIV-1 RNA was ≥400 copies/mL. Data for participants with respective gene mutation category has been reported. Participants with more than one mutation are counted more than once.
Time Frame: 48 weeks
Population: The FAS consisted of all participants who received at least 1 dose of study drug. "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
Number analyzed (Participants) | 3 | 4 | 3 | 13
participants
  With valid on-treatment results | 2 | 4 | 3 | 11
  PI Minor L10L/F | 0 | 0 | 0 | 1
  PI Minor L89L/I/M | 0 | 0 | 0 | 1
  PI Minor V77V/I | 0 | 0 | 0 | 1
  NNRTI K103K/N | 0 | 1 | 0 | 0
  NNRTI K103N | 0 | 0 | 1 | 1
  NRTI M184V | 0 | 0 | 1 | 0
  PI Minor K20K/R | 0 | 0 | 2 | 0
  Total with emergence | 0 | 1 | 3 | 4

19. Secondary Outcome: Percentage of Participants With Optimized Background Treatment Susceptibility Scores
Description: Data was summarized by the total ARV activity of the background regimen using simple and weighted total optimized background treatment susceptibility scores as well as by screening genotype. Simple total optimized background treatment (OBT) susceptibility scores were categorized as 0, 1, >=2 and weighted total OBT susceptibility scores were categorized as 0 to 0.5, 1 to 1.5 and >=2. However, net susceptibility scores were imputed for simple analysis based on genotype. Susceptibility scores indicate the level resistance to the study medication. Scores ranged from 0 to 1 as 1 = susceptible and potential low-level resistance; 0.5 = low and intermediate-level resistance; 0 = high-level resistance, where higher scores indicated lower resistance.
Time Frame: 48 weeks
Population: The FAS consisted of all participants who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Groups:
- Response: Participants with plasma HIV-1 RNA <48 copies/mL
- PDVF: Participants who meet the protocol-defined virologic failure
- Other Failure/Remainder: Participants with other failures
Arm/Group | Response | PDVF | Other Failure/Remainder
Number analyzed (Participants) | 49 | 23 | 31
Percentage of participants
  Simple score 0 | 0 | 0 | 0
  Simple score 1.0 | 8.2 | 4.3 | 0
  Simple score >=2.0 | 81.6 | 95.7 | 96.8
  Weighted score 0-0.5 | 6.1 | 30.4 | 29.0
  Weighted score 1.0-1.5 | 53.1 | 65.2 | 29.0
  Weighted score >=2.0 | 28.6 | 4.3 | 38.7

ADVERSE EVENTS:
Time Frame: Baseline up to 5 years
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | >=2 - <6 Years of Age, MVC Liquid Formulation | >=6 - <12 Years of Age, MVC Tablet Formulation | >=6 - <12 Years of Age, MVC Liquid Formulation | >=12 - <18 Years of Age, MVC Tablet Formulation
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/31 | 0/13 | 1/43
Serious Adverse Events (participants affected / at risk) | 5/16 | 5/31 | 3/13 | 10/43
Other Adverse Events (participants affected / at risk) | 12/16 | 25/31 | 10/13 | 34/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | >=2 - <6 Years of Age, MVC Liquid Formulation (N=16) | >=6 - <12 Years of Age, MVC Tablet Formulation (N=31) | >=6 - <12 Years of Age, MVC Liquid Formulation (N=13) | >=12 - <18 Years of Age, MVC Tablet Formulation (N=43)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Gastric fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Abscess oral (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 2
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | >=2 - <6 Years of Age, MVC Liquid Formulation (N=16) | >=6 - <12 Years of Age, MVC Tablet Formulation (N=31) | >=6 - <12 Years of Age, MVC Liquid Formulation (N=13) | >=12 - <18 Years of Age, MVC Tablet Formulation (N=43)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 5
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Conjunctival pallor (Eye disorders) | 0 | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 2 | 0 | 1
Hypermetropia (Eye disorders) | 0 | 0 | 0 | 1
Refraction disorder (Eye disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 4
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal pruritus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 2
Dental caries (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 7 | 3 | 4 | 9
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 5
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Salivary gland mucocoele (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Tongue disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 6 | 8 | 3 | 4
Asthenia (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 2 | 5
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Allergy to arthropod bite (Immune system disorders) | 0 | 1 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 0 | 2
Acarodermatitis (Infections and infestations) | 0 | 1 | 0 | 0
Bacterial vaginosis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 3 | 0 | 7
Bullous impetigo (Infections and infestations) | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 2 | 2 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 1 | 1 | 0 | 1
Fungal skin infection (Infections and infestations) | 1 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 0 | 2 | 2
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 0 | 0 | 1
Herpes virus infection (Infections and infestations) | 1 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0
Impetigo (Infections and infestations) | 1 | 1 | 0 | 1
Influenza (Infections and infestations) | 2 | 6 | 3 | 5
Latent tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Lice infestation (Infections and infestations) | 0 | 2 | 0 | 1
Nasopharyngitis (Infections and infestations) | 4 | 4 | 0 | 3
Oral herpes (Infections and infestations) | 1 | 2 | 0 | 1
Otitis externa (Infections and infestations) | 1 | 0 | 0 | 2
Otitis media (Infections and infestations) | 6 | 1 | 1 | 0
Otitis media acute (Infections and infestations) | 2 | 2 | 0 | 0
Otitis media chronic (Infections and infestations) | 2 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 1 | 0
Parotitis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 1 | 0 | 2
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 3 | 0 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 3 | 1 | 0 | 3
Sinobronchitis (Infections and infestations) | 0 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 1
Tinea capitis (Infections and infestations) | 2 | 1 | 0 | 0
Tinea faciei (Infections and infestations) | 0 | 1 | 0 | 0
Tinea infection (Infections and infestations) | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 2 | 0 | 2
Tooth abscess (Infections and infestations) | 0 | 0 | 1 | 0
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 6 | 2 | 5
Varicella (Infections and infestations) | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 3 | 2 | 3 | 1
Vulvovaginitis (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 2
Accidental exposure to product (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Underdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood HIV RNA increased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 1 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 2
Viral load increased (Investigations) | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Insulin resistance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 3
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 2 | 6
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 2
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 2
Hallucination (Psychiatric disorders) | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 1 | 0
Panic disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Breast enlargement (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 2 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acanthosis nigricans (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 1 | 1 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Conjunctivitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0 | 0
Viral rash (Infections and infestations) | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Traumatic ulcer (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1 | 0 | 0
Flat affect (Psychiatric disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Angular cheilitis (Infections and infestations) | 0 | 0 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Intellectual disability (Nervous system disorders) | 1 | 0 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study participating sites. Investigator may not disclose previously undisclosed confidential other than study results.